CLINICAL TRIAL: NCT01453751
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Intravenously in Patients With Type II Diabetes
Brief Title: Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered in Patients With Type II Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company dissolved
Sponsor: Ageless Regenerative Institute (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AD-US-DM2-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus Type II
Keywords: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Lipectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravenous Injection of AD-SVF (Experimental): Intravenous administration of AD-SVF.
  Interventions: Procedure: Harvesting and Implantation of Adipose-Derived Stromal Vascular Fraction (AD-SVF)

INTERVENTIONS:
Procedure: Harvesting and Implantation of Adipose-Derived Stromal Vascular Fraction (AD-SVF) — ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells.
  Other Names: Lipoaspiration; Liposuction

SUMMARY:
This will be an open-label, non-randomized, multi-center, patient sponsored study of Adipose-Derived Stromal vascular fraction cells implantation via intravenous infusion.

The intent of this clinical study is to answer the questions: 1) Is the proposed treatment safe and 2) Is treatment effective in improving the disease pathology of patients with diagnosed Type II Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Type 2 diabetes mellitus (as guideline WHO, 1999);
* Body mass index (BMI)≤35㎏/㎡;
* Fast blood glucose (FBG)≥7.0 mmol/L, and Hemoglobin A1c (HgbA1c)≥7％;
* Up to date on all age and gender appropriate cancer screening per American Cancer Society.

Exclusion Criteria:

* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. If patients have tested positive, they will be consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg or >180mmHg
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of insulin requirement by > 50% | 3 months and 6 months
Number of adverse events reported | up to the 6-month period following treatment
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.

SECONDARY OUTCOMES:
Improvement of Hemoglobin A1c(HbA1c) levels as compared to baseline | 3 months and 6 months
  Blood sample
reduction in requirement of insulin dosage compared to baseline | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon McQuillan, MD, Principal Investigator — Ageless Regenerative Institute
Locations (1):
- Ageless Regenerative Institute LLC, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided